CLINICAL TRIAL: NCT05222854
Title: Comprehensive Genomic Profiling Combined With Real Life Data of "The German-Registry of Incidental Gallbladder Carcinoma" the CONGENIAL Analysis Sub-study of the GR
Brief Title: Comprehensive Genomic Profiling Combined With Real Life Data of "The German-Registry of Incidental Gallbladder Carcinoma"
Status: Active, not recruiting | Type: Observational
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Other Study IDs: CONGENIAL
Record Dates: First submitted 2021-12-22; First posted 2022-02-03 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gallbladder Carcinoma
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — archival tumor tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter German- Registry of Incidental Gallbladder Carcinoma combining clinical real-world data and comprehensive genomic profiling. The registry collects medical data from clinical observation and molecular data derived from archival tumor tissue samples but does not define any medical intervention nor does it evaluate the efficacy or safety of the treatment decision made by the investigator.

DETAILED DESCRIPTION:
In the largest cohort of IGBC patients ever analysed in such a comprehensive approach

* determine the course of patients in this rare kind of cancer
* combine cGP analysis of histological tumor samples with clinical real-life data to get a comprehensive overview on IGBC patients analysed and evaluate data to identify possible further (targeted) treatment possibilities
* analyze potential risk factors associated with gallbladder carcinoma
* assess the frequency of targetable mutations in IGBC

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of incidental gallbladder carcinoma

* Patient ≥ 18 years old
* Patient already deceased
* Available tumor tissue (FFPE block)

Exclusion Criteria:

Patient under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients with gallbladder carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2099-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | Through study completion, an average of 2 years
  Overall Survival is defined as the time from date of first surgery, to the date of death (due to any cause).
proportion of patients with genomic alterations | Through study completion, an average of 2 years
  The primary outcome variable of the molecular sub-project is the proportion of patients with actionable genomic alterations, defined as number of patients with actionable mutations divided by the number of patients with completed F1 CDx testing. Additionally, the two-sided 95% exact confidence interval (Clopper-Pearson) will be given.

SECONDARY OUTCOMES:
The proportion of patients with actionable genomic alterations in all patients | Through study completion, an average of 2 years
  The proportion of patients with actionable genomic alterations in all patients, including those where no FoundationOne CDx test result may be obtained ± 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Götze, Prof., Principal Investigator — Institute of clinical cancer research
Locations (1):
- Frankfurter Institut für Klinische Krebsforschung IKF GmbH, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No